CLINICAL TRIAL: NCT03095365
Title: Dry Needling and Pain Neuroscience Education in Chronic Pain Patients
Brief Title: Dry Needling and Pain Education in the Treatment of Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, PhD, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03/2017
Record Dates: First submitted 2017-03-14; First posted 2017-03-29 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Pain, Neck
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dry needling (Active Comparator): Received Dry needling in the neck muscles.
  Interventions: Other: Dry needling
- Conventional treatment (Active Comparator): the participants received the conventional treatment for non-specific neck pain.
  Interventions: Other: Conventional treatment
- Dry needling and pain neuroscience education (Experimental): Received the same treatment as dry needling group and pain education.
  Interventions: Other: Dry needling; Other: Pain neuroscience education

INTERVENTIONS:
Other: Dry needling — Insertion of solid filament needles in the muscle
  Arms: Dry needling; Dry needling and pain neuroscience education
Other: Pain neuroscience education — Explanation of the functioning of the central nervous system, the differences between acute pain and chronic pain and the importance of thoughts and beliefs in the processing and chronification of pain
  Arms: Dry needling and pain neuroscience education
Other: Conventional treatment — Electrotherapy: Transcutaneous electrical nerve stimulation and microwaves
  Arms: Conventional treatment

SUMMARY:
to compare the effects on pain, disability and psychological factors of the combination of MTrP dry needling and pain neuroscience education to MTrPs dry needing alone and control electrotherapy usual care in patients with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical neck pain for at least 12 weeks
* 10% or higher on the Neck Disability Index questionnaire
* 20mm or higher on the Visual Analogue Scale (VAS) of neck pain
* Presence of at least one active myofascial trigger point

Exclusion Criteria:

* Neck pain associated with whiplash injuries
* Medical red flag history (i.e., tumour, fracture, metabolic diseases, rheumatoid arthritis, osteoporosis)
* Neck pain with cervical radiculopathy
* Neck pain associated with externalized cervical disc herniation
* Fibromyalgia syndrome
* Previous neck surgery
* Neck pain accompanied by vertigo caused by vertebrobasilar insufficiency or accompanied by non-cervicogenic headaches

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-05 (Actual)

PRIMARY OUTCOMES:
Pain using Visual Analogue Scale | 3 months
  Visual Analogue Scale: consists of a line of 100mm which represents the "no pain" on the left side of the same and the "worst pain imaginable" on the right side

SECONDARY OUTCOMES:
Medication intake | 3 months
  Medication use: number of pills
Disability using Neck Disability Index | 3 months
  Neck disability index: patients ability to function in daily life activities.
Kinesiophobia using Tampa Scale of Kinesiophobia | 3 months
  Tampa Scale of Kinesiophobia: participants pain-related fear of movement and (re)injury
Catastrophizing using Pain Catastrophizing Scale | 3 months
  Pain Catastrophizing Scale: propensity to catastrophize about pain
Pain anxiety using Pain Anxiety Symptoms Scale | 3 months
  Pain Anxiety Symptoms Scale: The anxiety behaviors associated with pain
Beck Depression Inventory-II | 3 months
  Self-report measure to assess the severity of depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Josue Fernandez-Carnero, PhD, Study Director — Universidad Rey Juan Carlos
Locations (1):
- Hospital Universitario Infanta Sofia, San Sebastián de los Reyes, Madrid, Spain

REFERENCES:
- [Derived] Valiente-Castrillo P, Martin-Pintado-Zugasti A, Calvo-Lobo C, Beltran-Alacreu H, Fernandez-Carnero J. Effects of pain neuroscience education and dry needling for the management of patients with chronic myofascial neck pain: a randomized clinical trial. Acupunct Med. 2021 Apr;39(2):91-105. doi: 10.1177/0964528420920300. Epub 2020 May 5. PMID 32370545